CLINICAL TRIAL: NCT06375772
Title: A Randomized, Double-blind, Placebo-controlled Phase 2 Study Using the Rhinovirus Challenge Model to Investigate the Efficacy and Safety of 2-Deoxy-D-Glucose as Pre-exposure Prophylaxis
Brief Title: A Controlled Human Rhinovirus Infection Study of 2-Deoxy-D-Glucose in Healthy Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Re-calculated sample size
Sponsor: G.ST Antivirals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2-DG-02
Record Dates: First submitted 2024-04-08; First posted 2024-04-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Acute Nasopharyngitis
MeSH Terms: conditions — Common Cold | interventions — Deoxyglucose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Drug (Active Comparator): Each subject receives a multiple dose of a 3.5% 2-Deoxyglucose as nasal spray solution. The maximum daily dose is 56 mg/day if applied 4 times/day, over 7 days.
  Interventions: Drug: 2-Deoxy-D-glucose
- Placebo (Placebo Comparator): Each subject receives a multiple dose of placebo as nasal spray solution. The dose is corresponding to the amount of solution needed in the serum group.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 2-Deoxy-D-glucose — Intranasal administration
  Other Names: 2-Deoxyglucose; 2-DG
  Arms: Study Drug
Other: Placebo — Intranasal administration
  Arms: Placebo

SUMMARY:
2-DG-02 is a randomized, placebo-controlled, double-blind Phase 2 study to investigate the efficacy and safety of 2-Deoxy-D-Glucose as a pre-exposure prophylaxis using the rhinovirus challenge model in healthy study participants.

DETAILED DESCRIPTION:
2-DG-02 is a randomized, placebo-controlled, double-blind Phase 2 study using the rhinovirus challenge model in healthy study participants aged 18 to 64 years.

The primary objective is to confirm the efficacy of 2-DG compared to placebo for the prevention of rhinovirus-associated illness.

Secondary objectives are

* to evaluate the effect of 2-DG on the occurrence and course of rhinovirus infection
* to evaluate the effect of 2-DG on the severity of symptoms of rhinovirus infection
* to evaluate safety and tolerability of 2-DG administrated over 1 week in the presence of rhinovirus exposure
* to evaluate pharmacokinetics of 2-DG

  128 subjects, who have been pre-screened and found to be seronegative to rhinovirus type 39, are randomized 1:1 to either 2-DG (pre-exposure prophylaxis) or placebo the day prior to inoculation. Subjects receive 2-DG or placebo starting from the day prior to inoculation until 5 days post inoculation.

Interim safety and efficacy reviews are performed by a Safety Monitoring Committee.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects 18 to 64 (inclusive at screening) years of age.
* Women of childbearing potential and all males must practice effective contraception during the study and be willing and able to continue contraception until end of study.
* Signed informed consent form prior to any study-related procedures.

Exclusion Criteria:

* Active smoker or history of smoking > 5 pack years.
* Upper or lower respiratory tract infection or febrile illness
* Presence (at screening) of serum RV-39 neutralizing antibody titer at greater than one in four (1:4) dilution.
* Nasopharyngeal swab indicative for Influenza or SARS-CoV2 infection by rapid antigen test at baseline.
* Prior inoculation with a virus from the same virus family as the challenge virus.
* Any anatomic or neurologic abnormality impairing the gag reflex, or associated with an increased risk of aspiration, or any abnormality significantly altering the anatomy of the nose or nasopharynx in a substantial way that may interfere with the aims of the study and in particular any of the nasal assessments or viral challenge.
* Positive Hepatitis B surface antigen (HBsAg), Hepatitis C virus antibody (HCV Ab), or human immunodeficiency virus antibody (HIV Ab) at screening.
* Any confirmed or suspected disease or condition associated with immune system impairment, including auto-immune diseases, asplenia or recurrent severe infections.
* Active allergic rhinitis or hay fever.
* Medical history or active asthma or chronic obstructive pulmonary disease (COPD) or any other pulmonary disease deemed by the investigator to increase the risk of participating in the study.
* Active nasal disease, e.g., nasal polyposis, significant septal deviation, chronic rhinosinusitis, etc.
* Frequent epistaxis or nasal sinus surgery within 3 months before baseline.
* Females: Pregnant, breast-feeding or intentions to become pregnant during the study.
* Evidence or history of drug or alcohol abuse.
* Positive test for drugs of abuse at screening or prior to study drug administration.
* Use of any prescribed or non-prescribed medication (except for contraceptives, paracetamol) within 1 week or less than 5 half-lives (whichever is longer) prior to the first administration of investigational product.
* Use of any over the counter cold prophylaxis products including nasal sprays, C-vitamins, zinc or Echinacea within 2 weeks prior to the first administration of investigational product.
* Participation in an investigational medical product, vaccine or device study within 3 months or 5 half-lives prior to the study period (whichever is longer), or more than 4 times in the past year.
* Hypersensitivity/allergy to any of the investigational product ingredients.
* Individuals with close contact to at risk patient group (infants less than 3 years, the extremely elderly >80 years or infirm, pregnant women, patients with severe lung disease(e.g., asthma/cystic fibrosis (CF)/COPD), patients with primary or secondary immunodeficiencies or ongoing immunosuppressive therapy).
* Any clinically relevant abnormal history, physical finding, 12-lead safety ECG, vital signs, laboratory value at screening or any known factor that could interfere with the objectives of the trial or the safety of the volunteer. In the case of uncertain or questionable results, tests performed during screening may be repeated before inclusion to confirm eligibility or judged to be clinically irrelevant.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-13 (Actual)

PRIMARY OUTCOMES:
The difference in the rate of rhinovirus-associated illness between 2-DG and placebo | baseline until day 22
  Difference in the rate of symptomatic illness and laboratory-confirmed infection

SECONDARY OUTCOMES:
Number of infected subjects | baseline, days 2-22 after start of dosing
  Difference in the number of subjects with laboratory-confirmed infections. A laboratory-confirmed infection is identified either by isolating rhinovirus on at least one day after the virus challenge using qPCR or by a 4-fold increase in neutralizing antibody titer to RV-39 from acute (day -1) to convalescent sera (day 22) using the neutralizing assay.
Difference in percent of infected subjects | baseline, days 2-22 after start of dosing
  Difference in percentage of subjects with laboratory-confirmed infections. A laboratory-confirmed infection is identified either by isolating rhinovirus on at least one day after the virus challenge using qPCR or by a 4-fold increase in neutralizing antibody titer to RV-39 from acute (day -1) to convalescent sera (day 22) using the neutralizing assay.
Difference in percent of days virus positive | days 2-6
  Difference in the percentage of days with a positive virus load. A positive virus load is determined by isolating rhinovirus on at least one day following the virus challenge, either using qPCR or a TCID50 assay.
Difference in peak nasal virus load | days 2-6
  Virus load is confirmed by isolating rhinovirus on at least one day after the virus challenge, using either qPCR or a TCID50 assay.
Difference in AUC nasal virus load | days 2-6
  Difference in AUC log 10 nasal virus load. Virus load is confirmed by isolating rhinovirus on at least one day after the virus challenge, using either qPCR or a TCID50 assay.
Difference in Total Jackson Symptom Score | days 2-6 after start of dosing
  The difference of total Jackson Symptom Score (4 point-liters scales from 0 to 3) where a lower score means a better outcome.
Duration of illness | days 2-15 after start of dosing
  In study participants with RAI duration of illness is the time to the first day of the two consecutive days with a total symptom score ≤ 1 that occurs after the subject has met the symptom criteria for a RAI. A lower duration means a better outcome.
Difference in percent of days Jackson Symptom Score positive | days 2-6 after start of dosing
  Percentage of days with positive Jackson Symptom Score ( score >2), where a lower percentage means a better outcome compared to placebo.
Difference in Peak Jackson Symptom Score | days 2-6 after start of dosing
  The highest daily total of all patient-reported symptoms on the Jackson Cold Scale (4 point-liters scales from 0 to 3 where a lower score means a better outcome compared to placebo).
Difference in peak total WURSS-21 | days 2-6 after start of dosing
  The highest daily total of all patient-reported symptoms on the WURSS-21 questionnaire (8-point Likert scales from 0 to 7) where a lower score means a better outcome compared to placebo.
Difference in AUC total WURSS-21 | days 2-6 after start of dosing
  Difference in AUC total WURSS-21 based a score recorded through the WURSS-21 questionnaire (8-point Likert scales from 0 to 7) where lower score means a better outcome compared to placebo.
Occurrence of adverse events (AEs) and adverse drug-reactions (ADRs) | from screening (day -56) until end of study (day 22± 2) after start of dosing
  Number of AEs and ADRs assessed by type, frequency and severity graded as per Common Terminology Criteria for Adverse Events (CTCAE).
Biodistribution of multiple doses of 2-DG in plasma samples | baseline, days 6 and 22± 2 after start of dosing
  Analysis of 2-DG concentrations in plasma samples measured by LCMS (μg/ml).
Biodistribution of multiple doses of 2-DG in nasal wash samples | baseline, days 2-6 and day 22± 2 after start of dosing
  Analysis of 2-DG concentrations in nasal wash samples measured by LCMS (μg/ml).

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid de Visser-Kamerling, PhD, Principal Investigator — Centre for Human Drug Research
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No